CLINICAL TRIAL: NCT01818453
Title: Genetic Predictors of Response to a Computerized Self-help Program for Depression
Brief Title: Can Genetics Predict Treatment Response to a Computerized Self-help Program for Depression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Christopher G. Beevers, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-01-0025
Record Dates: First submitted 2013-02-20; First posted 2013-03-26 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder; Mood Disorders
Keywords: Mood Disorders; Depression; Genetics; Treatment response; Treatment study
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized self-help program for depression (Active Comparator): Participants will have access to a computerized self-help program for depression, called deprexis, for 8 weeks.
  Interventions: Behavioral: Computerized self-help program for depression
- Wait List Control (No Intervention): Participants randomly assigned to a "wait list control" condition will wait 8 weeks after assignment before they can access the deprexis program.

INTERVENTIONS:
Behavioral: Computerized self-help program for depression — For 8 weeks, participants will engage in a computerized self-help program for depression, called deprexis. This program consists of 10 content modules representing different psychotherapeutic approaches broadly consistent with a cognitive-behavioral perspective. Modules are organized as simulated dialogues in which the program explains and illustrates concepts and techniques, engages the user in exercises, and continuously asks users to respond by selecting from response options. Subsequent content is then tailored to the users' responses, resulting in a simulated conversational flow. Participants can access the self-help program as often as they would like and since it is self-guided, they will determine how often they access the material. Each module can be completed in 10 to 60 minutes, depending on the user's reading speed, interest, motivation, and individual path through the program.
  Arms: Computerized self-help program for depression

SUMMARY:
The goal of this project is to determine whether genetic information can be used to predict response to an internet-based treatment of depression. Several studies now indicate that completing an internet-based treatment for depression, called Deprexis, can significantly improve symptoms of depression. However, not everyone improves. The purpose of this study is to determine whether genetic profile can predict who is likely to improve.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Have reliable access to the internet (i.e., dialup or broadband access)
* Be willing to donate saliva for DNA research
* Have a current symptoms of depression
* Be stable on medication and/or therapy (i.e. no changes within 2 weeks of study entry)

Exclusion Criteria:

* Any diagnosis of a psychotic or bipolar disorder
* Meeting for alcohol/drug dependence in the past year
* Having current suicidal risk warranting crisis intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (Self-Report) (QIDS-SR-16) | Administred every 2 weeks while the participant is engaged in the online deprexis treatment program to measure depression symptom severity.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | The HAM-D will be completed during the pre- and post-treatment phone interviews to assess depression symptom severity.
Inventory of Depression and Anxiety Symptoms (IDAS) | The IDAS will be completed as part of the pre- and post-treatment questionnaires to assess for symptoms of depression and anxiety.
Psychiatric Diagnostic Screening Questionnaire (PDSQ) | The PDSQ will be completed as part of the pre- and post-treatment questionnaires to screen for the most common DSM-IV Axis I disorders..
Risky Families Questionnaire (RFQ) | The RFQ will be completed as part of the pre-treatment questionnaires to assess early familial experiences and the harshness of family climate.
Massachusetts General Hospital Antidepressant Treatment History Questionnaire (ATRQ) | The ATRQ will be administered as part of the pre-treatment questionnaires to evaluate psychotropic efficacy.
Sheehan Disability Scale (SDS) | The SDS will be completed as part of the pre- and post-treatment questionnaires to evaluate symptom-related disability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Beevers, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Beevers CG, Pearson R, Hoffman JS, Foulser AA, Shumake J, Meyer B. Effectiveness of an internet intervention (Deprexis) for depression in a united states adult sample: A parallel-group pragmatic randomized controlled trial. J Consult Clin Psychol. 2017 Apr;85(4):367-380. doi: 10.1037/ccp0000171. Epub 2017 Feb 23. PMID 28230390